CLINICAL TRIAL: NCT04922203
Title: Are the Non Technical Skills Taught to Residents in Anesthesiology During in Situ Simulation Sessions Transferred to Clinical Practice
Brief Title: Transfer of Non-technical Skills From Simulation to Clinical Practice
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Jean François Brichant (Other)
Responsible Party: Sponsor-Investigator, Jean François Brichant, Sponsor, University of Liege
Organization: University of Liege (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2018-71
Record Dates: First submitted 2021-06-04; First posted 2021-06-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: in Situ Simulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Anesthesiology residents do not receive any in situ simulation sessions during the observation period
- Simulation group (Experimental): Anesthesiology residents receive in situ simulations sessions during the observation period
  Interventions: Other: in Situ Simulation

INTERVENTIONS:
Other: in Situ Simulation — 2 sessions of in situ simulation with 4 crisis scenarios and debriefing focused on non technical skills
  Arms: Simulation group

SUMMARY:
Since 1988, simulation has been proposed as a teaching tool in Anesthesia. The simulation environment allows to teach learners non-technical skills which are a combination of cognitive, social, and personal resources complementary to procedural skills that contribute to an efficient and safe performance.

Non-technical skills traditionally used in Anesthesia are task management, situational awareness, teamwork and decision making. They can be indirectly measured with validated scales (e.g. Anesthesia Non-Technical Skills (ANTS) system). In addition to these basic skills, specific skills such as Anesthesia Crisis Resource Management (ACRM) are required when the patient presents a critical clinical situation.

Simulation, as proposed by Gaba, was initially practiced in centers specifically designed for this purpose. More recently, we have proposed the model of in situ simulation, i.e. in the usual workplace with the usual work team, as another option for the practice of simulation.

There are many theories about the transfer of learning. Transfer can be defined as what remains of the completed training that the learner actually uses, i.e. the final real effect.

Nevertheless, almost 30 years after the introduction of simulation in the training of anesthesiologists, data demonstrating the interest of this teaching in terms of transfer of learning of non-technical skills to clinical practice or benefits for patients are rare.

The main objective of this study is to evaluate the transfer of non-technical skills taught in a training program including in situ simulation to clinical practice by anesthesiology residents.

ELIGIBILITY:
Inclusion Criteria:

- Internship in the ambulatory surgery unit

Exclusion Criteria:

- Refusal to participate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-05-28 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
ANTS (Anesthesia non technical skills) score | Once a day for 5 consecutive days between the first and the 15th day after enrollment in the study
  15 items - From 1(poor) to 4 (good) for each item - Minimum 15 - Maximum 60
ANTS (Anesthesia non technical skills) score | Once a day for 5 consecutive days between the 30th and 45th day after enrollment
  15 items - From 1(poor) to 4 (good) for each item - Minimum 15 - Maximum 60
ANTS (Anesthesia non technical skills) score | Once a day for 5 consecutive days between the 3rd and the 4th month after enrollment
  15 items - From 1(poor) to 4 (good) for each item - Minimum 15 - Maximum 60

SECONDARY OUTCOMES:
DOPS (Direct Observation of Procedural Skills) scale | Once within the first 15 days of enrollment
DOPS (Direct Observation of Procedural Skills) scale | Once between the 30th and the 45th day after enrollment
DOPS (Direct Observation of Procedural Skills) scale | Once between the 3rd and the 4th month after enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Liège - Sart-Tilman, Liège, Belgium